CLINICAL TRIAL: NCT00632801
Title: Does Chewing Gum After Elective Laparoscopic Colectomy Surgery Decrease Ileus?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in procedure nd medication used instead of gum
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Melanie Kalman, Melanie Kalman, PI, State University of New York - Upstate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 5579
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Ileus
Keywords: elective laparoscopic colectomy; chewing gum; ileus; post-operative care; colectomy
MeSH Terms: conditions — Ileus | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): Chewing gum or not
  Interventions: Other: chewing gum

INTERVENTIONS:
Other: chewing gum — The patients in the gum chewing group (intervention group) will chew one stick of gum the first post-operative day, after the nasogastric tube is removed or if they patient does not have a nasogastric tube, with the head of bed elevated a minimum of 30 degrees for 30 minutes, three times a day at set intervals

SUMMARY:
The incidence of ileus after laparoscopic colectomy continues to pose complications for the patient, staff, and the healthcare system. Postoperative ileus remains a source of morbidity and a major determinant of length of stay after abdominal surgery. Clinicians have devised strategies that minimize postoperative ileus. Gum chewing, an inexpensive intervention, is theorized to activate the cephalic- vagal reflex and increase the production of gastrointestinal hormones associated with bowel motility. Four studies examining gum chewing as an intervention to prevent ileus were found. These relatively few studies have demonstrated inconsistencies. Because of the small sample size of the four studies and the inconsistencies of the results, there is not enough evidence to change practice. There are no indications of risks associated with gum chewing as an adjunct therapy along with standard postoperative interventions. The purpose of this prospective, randomized control study is to examine if chewing gum in adult patients after elective laparoscopic colectomy decreases ileus compared with standard post-operative care.

Patients will be randomized by weeks admitted and the patients in the gum chewing group (intervention group) will chew one stick of gum the first post-operative day, after the nasogastric tube is removed or if they patient does not have a nasogastric tube, with the head of bed elevated a minimum of 30 degrees for 30 minutes, three times a day at set intervals: 0900, 1400, and 2100. The gum will be kept in the Accudose cabinet and distributed by the medication nurse. The gum chewing regimen will continue until the first bowel movement. All patients in the non-intervention group will receive standard preoperative and postoperative regimens.

Patient demographics that will be collected include gender, age, current medical condition, pre-operative medications, type of surgery, operative duration in minutes, anesthesia duration in minutes, estimated operative blood loss, whether they had an epidural or a PCA, date and time nasogastric tube was discontinued, length of stay, date of discharge, complications, and whether or not they had an ileus. Patients (if appropriate) and nurses will be instructed on how to complete the bedside bowel record to the nearest hour.

DETAILED DESCRIPTION:
Postoperative ileus remains a source of morbidity and a major determinant of length of stay after abdominal surgery. This unfortunate complication may certainly affect patient's satisfaction with their postoperative course. The postoperative care of a laparoscopic colectomy patient includes interventions that are evidence-based. Despite the evidence-based interventions, the incidence of ileus after laparoscopic colectomy continues to pose complications for the patient, staff, and the healthcare system. In the time period from January 1, 2006 to November 30, 2006 there were a total of 172 laparoscopic colectomies at St. Joseph's Hospital and 28 patients developed an ileus. Six percent of colectomy patients' recovery was altered by a prolonged ileus. This is comparably and slightly less then the National Veterans Affairs Surgical Quality Improvement Program's data for postoperative ileus of 7.5 % (Longo et al. 2000). However, the length of stay for patients with an ileus was 8.4 days greater then non ileus patients, with a significant increased cost per ileus patient of $15,422.86. Clinicians have devised strategies that minimize postoperative ileus. Adjunct therapies such as motility agents, early postoperative feeding regimens, and physical therapy have been tested in clinical trials, but are not routinely used because of their limited clinical efficacy (Matros, et al. 2006). Gum chewing, an inexpensive intervention, is theorized to activate the cephalic- vagal reflex, which is usually activated by food, and to increase the production of gastrointestinal hormones associated with bowel motility (Asao, et al, 2002).

Four studies examining gum chewing as an intervention to prevent ileus were found. These relatively few studies with a sample of postoperative abdominal surgical patients have demonstrated inconsistencies. Two studies found that the chewing gum group passed flatus and had a bowel movement sooner than the control group. One of these studies found a decreased length of stay. Two other randomized control studies found no statistical significance between the gum chewing and control groups as far as post-operative ileus or length of stay. Because of the small sample size of the four studies and the inconsistencies of the results, there is not enough evidence to change practice. The inexpensive method of gum chewing may be useful to decrease ileus in post-operative colectomy patients, which will decrease costs and length of stay. It could also decrease pain, emesis, and morbidity for patients. There are no indications of risks associated with gum chewing as an adjunct therapy along with standard postoperative interventions.

SPECIFIC OBJECTIVES: In adult elective laparoscopic colectomy patients does chewing gum decrease ileus compared with standard post-operative care? STUDY DESIGN: A prospective, randomized control design

SUBJECT SELECTION: (Include inclusion/exclusion criteria) All participants will be recruited at St. Joseph's Hospital. The sample will consist of all patients who are 18 years of age and older and are identified as adults on admission, and/or pre-admission for elective laparoscopic colectomy surgery. Inclusion criteria consist of all patients admitted to one surgical unit (3-1) from November 1, 2007 to August 1, 2008 with a non- emergent laparoscopic colectomy. Exclusion criteria consist of all patients with a history of metastatic disease, history of inflammatory bowel disease, abdominal radiation treatment, mint allergy (the gum is mint flavored), dentures, nasogastric tube drainage beyond the first postoperative morning, more then one bowel anastomosis during this surgery, conversion to pen colectomy, or admission to an ICI post-operatively.

STATISTICAL METHODS, DATA ANALYSIS AND INTERPRETATION: (Include the factors considered in determining an appropriate sample size) Data will be analyzed statistically. Descriptive statistics will be used to describe the entire sample, appropriate to the level of measurement of each. Independent t-tests for variables measured at ordinal or interval/ratio levels and chi-square for dichotomous variables will be used to compare the two groups on all demographic variables, hours since first flatus, and first bowel movement Analysis of co-variance may be used to statistically control for medical conditions found in the sample that were not excluded but could affect the findings.

STUDY PROCEDURES: (Describe all study methods chronologically. Distinguish clearly between treatment-related (standard care) and study-related procedures the subject will undergo).

NOTE: If the proposal includes genetic testing, some information about the genetic testing must be included. Please provide the following: 1. The type of study planned, 2. What genes are the investigators looking for, if known, 3. Why the genetic testing is being done (i.e., how it is relevant to the overall protocol), and 4. Where the work will be done.

After approval from St Joseph's IRB and SUNY Upstate's IRB, elective laparoscopic colectomy patients will be identified by the participating surgeons. At the time of preoperative instructions, a letter will be given or sent to the identified patient explaining the study (Appendix C). The day of pre-admission testing, the patient will be contacted by a study team member to review the study and will be asked to participate. If they agree, consent will be signed and the subjects will be assigned a number to ensure confidentiality.

The sample size of 50 will be randomized in block format, utilizing the weeks by number. The 38 weeks will be placed in a box; the first 19 weeks selected will be the gum chewing group, the second 19 weeks selected will be the non chewing group.

Each participant in the study will be educated to report to the nurse or self report on the bed side bowel report sheet the exact time to the hour that flatus is passed and the first bowel movement. The nursing staff on 3-1 will be instructed and monitored about documentation of gum chewing, first flatus to the nearest hour, and first bowel movement to the nearest hour. The data collection form will be completed. The length of the patients stay will be generated on discharge.

The patients in the gum chewing group (intervention group) will chew one stick of gum the first post-operative day, after the nasogastric tube is removed or if they patient does not have a nasogastric tube, with the head of bed elevated a minimum of 30 degrees for 30 minutes, three times a day at set intervals: 0900, 1400, and 2100. Sugar-free gum was used in all previous studies. Therefore, sugar free gum (Orbit Spearmint Sugarless Gum) will be used in this study. The gum will be kept in the Accudose cabinet and distributed by the medication nurse. The gum chewing regimen will continue until the first bowel movement. All patients in the non-intervention group will receive the standard preoperative and postoperative regimens. Patient demographics that will be collected include gender, age, current medical condition, pre-operative medications, type of surgery, operative duration in minutes, time left OR, anesthesia duration in minutes, estimated operative blood loss, whether the patient had an epidural or a PCA, date and time nasogastric tube was discontinued, length of stay, date of discharge, complications, and post-operative ileus. Patients and nurses will be instructed on how to complete the bedside bowel record to the nearest hour.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to one surgical unit (3-1) from November 1, 2007 to August 1, 2008 with a non- emergent laparoscopic colectomy.

Exclusion Criteria:

All patients with:

* History of metastatic disease
* History of inflammatory bowel disease
* Abdominal radiation treatment
* Mint allergy (the gum is mint flavored)
* Dentures
* Nasogastric tube drainage beyond the first postoperative morning
* More than one bowel anastomosis during this surgery
* Conversion to pen colectomy
* Admission to an ICI post-operatively.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Decrease ileus with intervention compared to standard post op care | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Kalmanm, RN PhD, Principal Investigator — SUNY UMU
Locations (1):
- SUNY UMU, Syracuse, New York, United States